CLINICAL TRIAL: NCT06490718
Title: Quality of Recovery After Major Breast Cancer Surgery: a Prospective Multicentre Randomized Triple Blinded Trial Comparing Erector Spinae Plane Block and Intravenous Lidocaine Infusion
Brief Title: Comparing Quality of Recovery Between ESPB and IV Lidocaine After Major Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CREC 2024.055-T
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-04

CONDITIONS: Breast Neoplasms
Keywords: Erector spinae plane block; Intravenous lidocaine infusion; Breast cancer surgery; Quality of recovery
MeSH Terms: conditions — Breast Neoplasms | interventions — Infusions, Intravenous

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized, triple-blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group ESPB (Active Comparator): For USG ESPB, 25 ml of 0.5% ropivacaine with 1:200,000 adrenaline will be drawn in a 25 ml syringe with a sterile label (available in a sterile package) displaying 'study drug for ESPB'.
  For IV infusion, 30 ml 0.9% saline will be drawn in a 50 ml syringe with a sterile label displaying 'study drug for IVI'. Both these syringes will be stored under strict aseptic precautions in a sterile tray until administration.
  Interventions: Drug: USG ESPB
- Group IVLI (Experimental): For USG ESPB, 25 ml of 0.9% saline will be drawn in a 25 ml syringe with a sterile label (available in a sterile package) displaying 'study drug for ESPB'.
  For IV infusion, 30 ml 2% lidocaine will be drawn in a 50 ml syringe with a sterile label displaying 'study drug for IVI'. Both these syringes will be stored under strict aseptic precautions in a sterile tray until administration. The 30 ml volume for 2% lidocaine is decided as it can cover for a 70kg patient for a 3-hour surgical period.
  Interventions: Drug: Intravenous Infusion

INTERVENTIONS:
Drug: USG ESPB — After obtaining the appropriate sonographic window, under strict aseptic precautions, the block needle is inserted in the plane of the US beam in a caudad to cranial direction until the tip is in contact with the transverse process (TP) at its lateral aspect. A test bolus of 0.9% saline (1-2 ml) is injected and sonographic evidence of erector spinae muscle displacement (posterior) from the underlying TP is sought to ensure that the tip of the block needle is indeed at the erector spinae muscle plane. The study drug from the 25 ml syringe with the label 'study drug for ESPB' (containing either 25 ml of 0.5% ropivacaine with 1:200,000 adrenaline or 0.9% saline depending on the group allocation) is injected in small aliquots over a minute. The anaesthesiologist performing the block and the patient is blinded to the group allocation.
  Successful injection reveals a clearly delineated posterior displacement of the erector spinae muscle.
  Arms: Group ESPB
Drug: Intravenous Infusion — Following ultrasound-guided erector spinae plane block (USG ESPB), patients will be transferred to the operating room. General anesthesia (GA) will be administered according to a standardized protocol.
  Study Drug Infusion:
  Immediately after securing the airway, an intravenous infusion from a 50 ml syringe labeled "study drug for IVI" will commence. The study drug contains either 30 ml of 2% lidocaine or 0.9% saline, depending on group allocation. The infusion begins with a bolus rate of 0.1 ml/kg over 10 minutes and continues at 0.1 ml/kg/hr until surgical wound closure.
  Arms: Group IVLI

SUMMARY:
The erector spinae plane block (ESPB) is gaining popularity as a regional anesthetic technique for major breast cancer surgery. Although there is controversy about its mechanism of action, emerging evidence suggests that clinical analgesia observed after ESPB in breast surgery may be due to rapid and sustained local anesthetic absorption from the injection site. Hence intravenous LA infusion (IVLI) during the perioperative period could offer an effective alternative to invasive ESPB.

DETAILED DESCRIPTION:
Major Breast Cancer Surgery (BCS), including mastectomy or modified radical mastectomy (MRM), is a globally prevalent procedure. Unfortunately, it is associated not only with significant acute postoperative pain but also a high incidence of chronic postsurgical pain (30-50%) . To improve outcomes, regional anesthetic techniques have been explored, including thoracic paravertebral block (TPVB) and ultrasound-guided erector spinae plane block (ESPB). While TPVB is considered the gold standard, it carries potential complications such as pleural puncture and pneumothorax. In contrast, ultrasound-guided (USG) ESPB is gaining popularity due to its technical simplicity and safety. However, controversy surrounds its mechanism of action, particularly the variable cutaneous sensory loss over anterior thoracic dermatomes. An emerging theory suggests that ESPB's clinical analgesia results from rapid and sustained local anesthetic (LA) absorption from the injection site. As an alternative, intravenous LA infusion (IVLI) during the perioperative period may offer equivalent analgesia without the invasiveness of ESPB. IV lidocaine, known for its substantial analgesic properties, persists beyond its typical duration of action, likely through mechanisms beyond sodium channel blockade. Although IV lidocaine has been established as part of multimodal analgesia in various perioperative settings, data specific to major BCS remain scarce. In this prospective, multicenter, randomized, triple-blind trial, the investigators aim to compare quality of recovery (assessed using the validated Quality of Recovery 15 [QoR15] score) between USG ESPB and IVLI. The investigator's hypothesis is that the quality of recovery after major breast cancer surgery with IVLI will be comparable to that achieved with USG ESPB.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* 18 to 75 years of age
* Patients scheduled for primary breast cancer surgery-mastectomy, modified radical mastectomy and breast conservation surgery with sentinel lymph node biopsy +/- axillary dissection will be included in this study.

Exclusion Criteria:

* Patient refusal,
* Local skin site infection,
* Coagulopathy,
* History of allergy to local anaesthetics, and
* Patients with hepatic, renal and cardiac dysfunction

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery | At 24 hours post surgery
  Quality of Recovery-15: a minimum score of 0 (poor recovery) and a maximum score of 150 (excellent recovery)
Area under the curve of postoperative pain | Over the first 24 hours post surgery
  Area under the curve of postoperative pain numerical rating score at rest and movement

SECONDARY OUTCOMES:
Postoperative opioid consumption | At 24 and 48 hour post surgery
  Total postoperative morphine equivalent consumption

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, FRCA, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- The First Affiliated Hospital, Guangzhou, Guangdong, China
- North District Hospital, Sheung Shui, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided